CLINICAL TRIAL: NCT04945811
Title: Role of Interleukin-6 and Procalcitonin in Evaluating COVID 19 Disease Severity - an Experience at CMH Quetta
Brief Title: Role of Interleukin-6 and Procalcitonin as Novel Inflammatory Biomarkers in Evaluating COVID 19 Disease Severity - an Experience at CMH Quetta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FARAH AFZAL (Other)
Responsible Party: Sponsor-Investigator, FARAH AFZAL, CLASSIFIED SPECIALIST, Combined Military Hospital, Pakistan
Organization: Combined Military Hospital, Pakistan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMHQ3
Record Dates: First submitted 2021-06-29; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Covid19 Positive Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interlukein 6 and procalcitonin (Experimental): Interlukein 6 and procalcitonin levels in COVID 19 patients
  Interventions: Diagnostic Test: Interlukein 6 and procalcitonin serum levels

INTERVENTIONS:
Diagnostic Test: Interlukein 6 and procalcitonin serum levels — Blood tests

SUMMARY:
Serum Interleukin-6 and Procalcitonin of 100 consenting COVID 19 positive patients from April 2020 - May 2021 were assessed at Pathology department CMH Quetta and the results were correlated with severity of lung involvement on HRCT Chest

DETAILED DESCRIPTION:
Objective: To explore the relation between Interleukin-6 and Procalcitonin with COVID severity on HRCT Chest Study Design: Randomized Control Trial (Clinical Trials. gov Identifier: NCT04798391) Place and duration of study: Pathology, Radiology & ENT Department CMH Quetta from April 2020 - May 2021 Methodology: Serum Interleukin-6 and Procalcitonin of 100 consenting COVID 19 positive patients from April 2020 - May 2021 were assessed at Pathology department CMH Quetta and the results were correlated with severity of lung involvement on HRCT Chest Results: Serum Interlukin-6 levels were raised in 97 (97%) patients with mean levels of 20.43 + 19.66 (pg/ml). Serum procalcitonin levels were raised in 95 (95%) patients with mean levels of 0.4331 + 0.24 (ng/ml). A P value of <0.001 was calculated on Independent Sample T-test for both serum interlukin-6 and serum procalcitonin as correlated with severity of lung involvement on HRCT Chest.

Conclusion: Interlukin-6 and procalcitonin are excellent biomarkers for diagnosis and predicting severity of COVID19 pneumonia.

Keywords: Covid19 pneumonia, Interlukin-6, procalcitonin.

ELIGIBILITY:
Inclusion Criteria:

* positive PCR of COVID 19

Exclusion Criteria:

* NEGATIVE PCR of COVID 19

Ages: 38 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Levels of inflammatory biomarkers is raised in accordance with severity of COVID 19 | 2 days
  serum Interlukin-6 levels was measured on COBAS-e 411 Immunoassay analyzer using electro chemiluminescence methodology using Roche Interlukin-6 kit with raised levels taken as > 7 pico gram / milliliter (pg/ml). Serum procalcitonin were also measured by similar methodology using Roche procalcitonin kit with raised levels taken as > 0.15 nano gram / milliliter (ng/ml).
  COVID 19 pneumonia was categorized on HRCT chest as Mild with total score 7 or less, moderate with score from 8 - 17, and severe with score more than 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Cmh Quetta, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No